CLINICAL TRIAL: NCT03195920
Title: Feasibility Study of an Enhanced Lithotripsy System in the Treatment of Urinary Stone Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim data was sufficient for study purpose
Sponsor: Avvio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-02
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Urinary Stone
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Single arm trial with the Enhanced Lithotripsy System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Enhanced Lithotripsy System (Experimental): Treatment for urinary stones with the Enhanced Lithotripsy System
  Interventions: Device: Enhanced Lithotripsy System

INTERVENTIONS:
Device: Enhanced Lithotripsy System — The Enhanced Lithotripsy System is a type of lithotripsy system comprising a console, treatment head, and Acoustic Energy Focusing material. Operation of the Enhanced Lithotripsy System entails combined action of extracorporeal insonation and Acoustic Energy Focusing material to fragment urinary stones.

SUMMARY:
This is a single arm, single center study to assess the safety and efficacy of a form of extracorporeal lithotripsy, called the Enhanced Lithotripsy System, to treat urinary stones.

DETAILED DESCRIPTION:
This is a single arm, single center study to assess the safety and efficacy of a form of extracorporeal lithotripsy, called the Enhanced Lithotripsy System, to treat urinary stones. Subjects will be treated up to 2 times with the Enhanced Lithotripsy System and followed for 30 days after the last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting with one urinary stone-apparent on a computed tomography scan within the last 14 days
* Males and females aged 18 or older
* Capable of giving informed consent, and willing to have the informed consent process videotaped
* Stone size, as estimated by pre-operative computed tomography, with all dimensions 15 mm or less.

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals with radiolucent stones
* Individuals with stones in the lower pole of kidney
* Individuals not following up in the treating hospital
* Individuals with history of cystinuria
* Individuals with urine pH below 5.5
* Individuals with untreated urinary tract infection
* Individuals who are not willing to use adequate method of contraception during the study period
* Women who are pregnant, lactating or planning pregnancy during the study period
* Individuals with a coagulation abnormality or taking prescription anticoagulants.
* Individuals with mobility issues who are unable to comfortably lie still for up to 30 minutes or roll from their back to their side
* Individuals belonging to a vulnerable group (pregnant, mentally disabled, physically disabled, prisoner, etc.)
* Individuals with a body mass index greater than 35
* Individuals with ASA score of 3 or greater general anesthesia risk level
* Known sensitivity to possible medications used before, during, or after the treatment procedure, including but not limited to the following: sedative agents, general anesthetics, topical anesthetics, and opioid analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with serious device-related adverse events (safety) | 30 days after last treatment session
  Safety: Proportion of subjects with serious device-related adverse events

SECONDARY OUTCOMES:
Successful treatment of urinary stone | 14 days after last treatment session
  Proportion of subjects with successful treatment or urinary stone

OTHER OUTCOMES:
Change in pain score | Baseline and Post Procedure Days 1, 2, 3, 7, 14, and 30
  Pelvic Pain of the Patient (Min - Zero, Max - 10), Higher score means more pain
Time to passage of stones | 30 days after last treatment session
  Post-Treatment time to passage of stone fragments after treatment
Pain medication usage | Baseline and Days 1, 2, 3, 7, 14, and 30
  Use and quantity of pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Desai, MS, FRCS, Principal Investigator — Muljibhai Patel Urological Hospital
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided